CLINICAL TRIAL: NCT01538719
Title: Randomized, Double-Blind, Placebo-Controlled Trial if IL1-TRAP, Rilonacept, in Systemic Sclerosis -A Phase I/II Biomarker Trial
Brief Title: IL1-TRAP, Rilonacept, in Systemic Sclerosis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Boston University (Other)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Robert Simms, Professor of Medicine, Boston University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H31332
Record Dates: First submitted 2012-02-21; First posted 2012-02-24 (Estimated); Results first posted 2018-05-01 (Actual); Last update posted 2018-05-01 (Actual); Status verified 2018-04

CONDITIONS: Scleroderma; Systemic Sclerosis; Diffuse Scleroderma; Diffuse Systemic Sclerosis
MeSH Terms: conditions — Scleroderma, Diffuse; Scleroderma, Systemic | interventions — rilonacept

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): 2:1 randomization
  Interventions: Other: Placebo
- Rilonacept (Active Comparator): 2:1 randomization
  Interventions: Drug: Rilonacept

INTERVENTIONS:
Drug: Rilonacept — Patients randomized to active study drug will receive Rilonacept 320 mg subcutaneously (SQ) on day 0 and 160 mg SQ each week for 5 additional weeks
  Other Names: IL1-TRAP
  Arms: Rilonacept
Other: Placebo — Patients randomized to placebo will receive saline subcutaneously (SQ) on day 0 and each week for 5 additional weeks
  Arms: Placebo

SUMMARY:
Scleroderma,also known as systemic sclerosis (SSc), is a multisystem disease affecting skin and other tissues including joints, muscles, lungs, the gastrointestinal tract and kidneys and tissue fibrosis is widespread. SSc presents special problems for developing therapies due to the heterogeneous clinical presentation, the variability of disease progression and the difficulty quantifying the extent of disease. For most disease manifestations, treatment is primarily symptomatic and generally inadequate.

This study will utilize a 4-gene biomarker of skin disease as the primary efficacy outcome in a short duration, placebo-controlled clinical trial of rilonacept, designed to provide preliminary data for a larger trial. These gene biomarkers should provide a strong surrogate for such trials in the future and, if IL-1 is indeed the cytokine leading to fibrosis in this disease, provide a highly significant start to finding a therapeutic for SSc that for the first time might dramatically affect fibrosis. A central hypothesis of this study is that IL-1 inhibition will downregulate the 4-gene biomarker over a relatively short period of time, much shorter than is historically thought necessary to see changes in the MRSS, a skin score measurement tool. Entry criteria will include the recent onset of diffuse cutaneous SSc as this is the population most likely to show progressive skin disease and also the population examined in previous studies showing correlations between MRSS and the 4-gene biomarker.

Secondary outcomes will include other validated measures of SSc disease activity. MRSS and SSc health assessment questionnaire (SHAQ), will be followed during the trial. This study will also test the effect of rilonacept on global skin gene expression using microarray analyses of skin biopsies. In addition, serum biomarkers of SSc disease activity (COMP, THS-1 and IFI44) and a biomarker of inflammasome activation (CRP) will be tested before and after treatment.

DETAILED DESCRIPTION:
Overview of Systemic Sclerosis

Scleroderma, also known as systemic sclerosis (SSc), is a multisystem disease affecting skin and, more variably, other tissues, commonly including joints, muscles, lungs, the gastrointestinal tract and kidneys. It is one of a group of diseases in which fibrosis is associated with organ dysfunction. Fibrosis can involve the liver (Lefton et al., 2009; Pinzani et al., 2005), lung(Frankel and Schwarz, 2009), kidneys (Schnaper, 2005), and less commonly other organs, representing a final common pathway to organ dysfunction. In SSc tissue fibrosis is widespread, variably involving skin, lungs and the gastrointestinal tract.

Although SSc can affect almost any part of the body, skin disease is the most consistent clinical manifestation. Skin disease typically starts in the hands with an edematous phase of hand swelling lasting one to several months. The skin then progressively thickens and tethers to underlying tissues. In diffuse cutaneous SSc (dcSSc), skin thickening, induration and tethering typically extend proximally up the arm and can involve the torso, abdomen, face and legs. Patients with limited cutaneous SSc (lcSSc) have skin disease limited to below the elbow and face and neck as well as other characteristic clinical features. SSc skin pathology (diffuse and limited cutaneous SSc) shows fibrosis and variable perivascular lymphocyte infiltration in the deep reticular dermis.

SSc affects multiple other body systems. Most severe complications are seen more frequently in dcSSc with considerable morbidity and mortality(Steen and Medsger, 2000). Lung disease manifests as interstitial fibrosis or pulmonary arterial hypertension (PAH, more common in lcSSc). Lung disease remains the leading cause of death among SSc patients. Gastrointestinal disease primarily results from dysmotility. In the esophagus and stomach this most commonly leads to esophagitis. In the small and large bowel this most commonly leads to constipation, bowel obstruction and/or malnutrition. Renal disease is primarily manifest as accelerated hypertension and renal insufficiency. Angiotension converting enzyme inhibitors are generally though not uniformly effective for treating this manifestation, which previously led to significant mortality.

Other important clinical manifestations include cold-induced vasospastic disease in extremities (Raynaud's phenomenon) and digital ulcers. SSc can also have cardiac manifestations. Pericarditis is the most frequent cardiac manifestation. Subclinical pericarditis is common with large effusions developing occasionally. Myocardial involvement with low-grade myocardial fibrosis is relatively common, but not frequently of clinical importance (Follansbee et al., 1985). Fibrosis most commonly manifests as the appearance of a septal infarction pattern on EKG in patients with normal coronary arteries, or as ventricular conduction delays. Occasionally myocardial fibrosis leads to heart failure. Cardiac arrhythmias are seen in ~5% of patients with SSc. Most common are atrial or ventricular ectopy, generally not associated with more serious rhythm disturbances. However, thallium perfusion defects are associated with sudden cardiac death (Steen et al., 1996).

Current treatment for SSc is limited (Steen, 2001). For most disease manifestations treatment is primarily symptomatic and generally inadequate. The exception is renal disease, scleroderma renal crisis, once a major cause of mortality in SSc patients, can often be treated successfully with angiotensin converting enzyme inhibitors. Pulmonary complications now represent the major cause of mortality. Cyclophosphamide provides some benefit in patients with interstitial lung disease (ILD), the most lethal complication of SSc. However, the effect of this agent on SSc-associated ILD is modest and transient (Tashkin et al., 2006; Tashkin et al., 2007). Pulmonary arterial hypertension (PAH) also leads to considerable mortality in SSc patients. PAH may respond to vasodilators such as epoprostanol and bosentan, but frequently responses are incomplete and mortality still high(Badesch et al., 2009) . Bowel hypomotility also leads to considerable morbidity and sometimes mortality. Esophageal hypomotility is treated, frequently without success, with pro-motility and acid-blocking agents. Dysmotility of the lower bowel and its complications are even more difficult to treat with pro-motility agents providing modest relief in some patients and antibiotics helping in cases of small bowel overgrowth. Thus there are limited therapeutic alternatives for SSc patients faced with progressive lung or bowel disease.

Skin fibrosis, the hallmark feature of SSc remains without effective treatment. Although skin changes in SSc are not a cause of mortality, they cause considerable morbidity, may reflect similar pathological processes to those that occur in the bowel and lungs, correlate highly with prognosis and disease progression in other organ systems, and can be reproducibly assessed by skin score testing. Skin disease is of particular interest for evaluation in clinical trials since it is easily biopsied and can thus be repeatedly assessed for pathological changes during clinical trials (Lafyatis et al., 2009).

Part of the difficulty in finding effective treatments for SSc has been a continuing uncertainty regarding what initiates pathogenesis. The cause of disease manifestations in SSc remains obscure, although three major pathophysiologic explanations have been advanced. Prominent pathologic changes in dermal and pulmonary tissues show fibrosis, suggesting abnormalities in matrix deposition. Vascular disease, resulting in scleroderma renal crisis, digital ischemia and pulmonary hypertension suggests dysfunction of the vascular endothelium. Autoantibodies in SSc patient sera suggest that immune dysfunction and autoimmunity may contribute to or cause disease. The different pathological features in different organs have provided support for each of these mechanisms, but not clarified which is most important in overall pathogenesis.

Background: IL-1 Rationale for blocking IL-1 in Systemic Sclerosis: The inflammasome and fibrosis Several observations have implicated IL-1 in fibrotic diseases and SSc. Environmental or occupational exposure to silica dust leads to fibrosis (Cohen et al., 2008) and has been associated with SSc (Rustin et al., 1990). Recently, several groups have shown in murine models that silica dust activates inflammation and fibrosis through the inflammasome (Cassel et al., 2008; Hornung et al., 2008) . Activation of the inflammasome also contributes to bleomycin-induced lung injury (Gasse et al., 2007).

Rilonacept blocks IL-1β signaling by acting as a soluble decoy receptor that binds IL-1β and prevents its interaction with cell surface receptors. Rilonacept also binds IL-1α and IL-1 receptor antagonist (IL-1ra) with reduced affinity.

Rationale for Rilonacept In This Study SSc presents special problems for developing therapies due to the heterogeneous clinical presentation, the variability of disease progression and the difficulty quantifying the extent of disease. The variability of disease progression presents particular challenges for deciding whom to treat, leading to overtreatment of patients as well as misinterpretation of open label trials. This heterogeneity of disease progression has also required recruitment of relatively large patient numbers into clinical trials, many with skin disease that is going to stabilize or improve spontaneously (Amjadi et al., 2009).

Purpose/Objectives

This study will utilize a 4-gene biomarker of skin disease as the primary efficacy outcome in a short duration, placebo-controlled clinical trial of rilonacept, designed to provide preliminary data for a larger trial. The change in 4-gene SSc biomarker skin score from day 0 to day 42 or last observation carried forward(LOCF) will be measured in both rilanocept-treated patients as well as placebo patients and the scores will be compared. These gene biomarkers should provide a strong surrogate for such trials in the future and, if IL-1 is indeed the cytokine leading to fibrosis in this disease, provide a highly significant start to finding a therapeutic for SSc that for the first time might dramatically affect fibrosis. A central hypothesis of this study is that IL-1 inhibition will downregulate the 4-gene biomarker over a relatively short period of time, much shorter than is historically thought necessary to see changes in the MRSS. Entry criteria will include the recent onset of dcSSc as this is the population most likely to show progressive skin disease and also the population examined in previous studies showing correlations between MRSS and the 4-gene biomarker.

Secondary outcomes will include other validated measures of SSc disease activity. MRSS, SSc health assessment questionnaire (SHAQ), which includes the health assessment questionnaire (HAQ) and a SSc specific, patient visual analogue scale (VAS) for organ specific involvement will be followed during the trial. Several studies suggest that the SHAQ accurately measures disease activity and may detect smaller changes in health status. This study will also test the effect of rilonacept on global skin gene expression using microarray analyses of skin biopsies. In addition, serum biomarkers of SSc disease activity (COMP, THS-1 and IFI44) and a biomarker of inflammasome activation (CRP) will be tested before and after treatment. The change in MRSS score, SHAQ score, skin myofibroblast score, gene expression, CRP and serum biomarkers from day 0 to day 52 will be compared between the rilanocept-treated patients and the placebo-treated patients.

ELIGIBILITY:
Inclusion Criteria:

* Must meet the American College of Rheumatology criteria for systemic sclerosis with diffuse cutaneous involvement and < 24 months since the onset of the first SSc manifestation other than Raynaud's phenomenon; or has had an increase of MRSS by 5 in the last 6 months.
* Must have a MRSS of ≥ 15.
* Male or female patients ≥ 18 years of age.
* Able and willing to give written informed consent and comply with the requirements of the study protocol.

Exclusion Criteria:

* Treatment with any investigational agent within 4 weeks of screening or 5 half-lives of the investigational drug (whichever is longer).
* Ongoing use of high dose steroids (> 10mg/day prednisone or equivalent) or unstable steroid dose in the past 4 weeks.
* Treatment with immunosuppressive (other than low dose steroids), cytotoxic or anti-fibrotic drug within 4 weeks of screening.
* The patient has positive viral hepatitis B, hepatitis C or HIV serologies on screening laboratories. (Patients with a positive hepatitis B surface antibody (HBsAb) test with a history of prior hepatitis B immunization are eligible as long as other criteria are met (i.e., negative tests for: hepatitis B surface antigen [HBsAg], hepatitis B core antibody [HBcAb], and hepatitis C virus antibody [HCVAb]).)
* Known active bacterial, viral fungal mycobacterial, or other infection (including tuberculosis or atypical mycobacterial disease, but excluding fungal infections of nail beds) or any major episode of infection requiring hospitalization or treatment with i.v. antibiotics within 4 weeks of screening.
* Patients must have a negative PPD tested within 6 months of the time of screening, or past positive PPD treated with appropriate antibiotic prophylaxis.
* Patients with a history of malignancy within the past 5 years.
* Moderate to severe hepatic impairment, i.e., Child-Pugh Class B or C.
* Scleroderma renal crisis within 6 months or creatinine greater than 2.0
* Pregnancy (a negative pregnancy test will be performed for all women of childbearing potential on study day 0 and 42).
* Male and female patients of child-producing potential must agree to use effective contraception while enrolled on study and receiving the experimental drug, and for at least 3 months after the last treatment.
* Nursing mothers
* Gastrointestinal involvement requiring total parenteral nutrition or hospitalization within the past 3 months for pseudo-obstruction
* Moderately severe pulmonary disease with FVC < 60%, or DLCO < 50% predicted.
* Moderately severe cardiac disease with either a history of significant arrhythmia (not to include conduction delays other than trifascicular block, or PVCs or PACs < 5/minute), clinically significant heart failure, or unstable angina.
* Hemoglobin: < 8.5 gm/dL
* White blood count < 3,000/mm3 or total neutrophil count < 1,500
* Platelets: < 100,000/mm3
* AST or ALT > 2.5 x Upper Limit of Normal.
* Total bilirubin > 1.5 x upper limit of normal (ULN). Patients with Gilbert's Disease may be included if their total bilirubin is ≤ 3.0 mg/dL.
* Patients should not have received any live vaccine within 30 days of trial entry
* Patients with a history of rilonacept allergy will be excluded.
* Patients who, in the opinion of the Investigator, have significant medical or psychosocial problems that warrant exclusion. Examples of significant problems include, but are not limited to:
* Other serious non-malignancy-associated medical conditions that may be expected to limit life expectancy or significantly increase the risk of SAEs.
* Any condition, psychiatric, substance abuse, or otherwise, that, in the opinion of the Investigator, would preclude informed consent, consistent follow-up, or compliance with any aspect of the study
* Current use of TNF-blockers within 4 weeks of screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2011-12 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-08-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert W Simms, MD, Principal Investigator — Boston University Medical Center-Rheum/Arthritis Center
Locations (1):
- Boston University Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Mantero JC, Kishore N, Ziemek J, Stifano G, Zammitti C, Khanna D, Gordon JK, Spiera R, Zhang Y, Simms RW, Lafyatis R. Randomised, double-blind, placebo-controlled trial of IL1-trap, rilonacept, in systemic sclerosis. A phase I/II biomarker trial. Clin Exp Rheumatol. 2018 Jul-Aug;36 Suppl 113(4):146-149. Epub 2018 Sep 30. PMID 30277862

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 2 subjects withdrew consent and 3 found to be ineligible, leaving 19 for randomization.
Period: Overall Study
Arm/Group | Placebo | Rilonacept
Started | 7 | 12
Completed | 5 | 12
Not Completed | 2 | 0
Not completed — Lost to Follow-up | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Rilonacept | Total
Number analyzed (Participants) | 7 | 12 | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.86 (11.10) | 51.33 (7.33) | 50.79 (8.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 7 | 9
  Male | 5 | 5 | 10
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 7 | 12 | 19

OUTCOME MEASURES:

1. Primary Outcome: Change in 2- Gene Biomarker
Description: To investigate the effect of rilonacept on 2-gene biomarker expression in skin after treatment with rilonacept compared to pre-treatment 2-gene biomarker expression. These were measured at visit 3 (Day 42) and visit 1 (Day 0). This was calculated using a previously validated equation (MRSS = -27.6844 + [4.46(baseline THBS1)] + [5.31(ΔMS4A4A) + 4.96(ΔTHBS1)]). In this equation the expression of two genes (THBS1 and MS4A4) in collected samples are measured via nanostring, and then the expression levels of each gene are inserted into the equation in order to obtain the 2- gene biomarker score. A high biomarker score is equivalent to a high skin score, suggesting a higher severity of the disease.
Time Frame: Visit 3 (Day 42) - Visit 1 (Day 0)
Population: Analysis run on 4 available samples in placebo arm.
Measure: Mean (95% Confidence Interval); unit: 2- gene biomarkers score
Arm/Group | Placebo | Rilonacept
Number analyzed (Participants) | 4 | 12
2- gene biomarkers score | -2.67 [-5.92 to 0.57] | 0.42 [-2.97 to 3.82]

2. Secondary Outcome: Change in Modified Rodnan Skin Score
Description: Change in Modified Rodnan Skin Score over time. The fully validated modified version of the Rodnan skin thickness score was used. On this scale, a total of 17 skin sites are evaluated, including the face, upper arms, forearms, dorsum of the hands, fingers, chest, abdomen, thighs, forearms and feet. The total score can range from 0 to 51, with higher scores indicating greater severity of skin thickening and involvement (MRSS-51). Each of the 17 skin sites are scored from 0 to 3, where the following criteria apply: 0, normal skin; 1, thickened skin; 2, thickened and unable to pinch; and 3, thickened and unable to move. Scores from visit 3 (Day 42) and visit 1 (Day 0) were compared.
Time Frame: Visit 3 (Day 42) - Visit 1 (Day 0)
Measure: Mean (Full Range); unit: Units on the Modified Rodnan Skin Score
Arm/Group | Placebo | Rilonacept
Number analyzed (Participants) | 7 | 12
Units on the Modified Rodnan Skin Score | -0.4 [-5 to 9] | -0.6667 [-5 to 14]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from screening (Day -28) up to study completion (visit 4 / Day 84)
Arm/Group | Placebo | Rilonacept
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/12
Other Adverse Events (participants affected / at risk) | 2/7 | 10/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=7) | Rilonacept (N=12)
Pain (Skin and subcutaneous tissue disorders) | 1 | 0
Allergic Reaction on Abdomen (Skin and subcutaneous tissue disorders) | 0 | 1
Digital Ulcer Worsening (Skin and subcutaneous tissue disorders) | 0 | 1
Abscess on Back (Skin and subcutaneous tissue disorders) | 0 | 1
Left Breast Swelling (Skin and subcutaneous tissue disorders) | 0 | 1
Malaise (General disorders) | 1 | 0
Injection Site Reaction (Skin and subcutaneous tissue disorders) | 0 | 2
Fatigue (General disorders) | 0 | 2
Infection (Skin and subcutaneous tissue disorders) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes